CLINICAL TRIAL: NCT04336358
Title: Telemedicine Versus Standard Care for First Trimester Abortion in South Africa: a Randomized Controlled Noninferiority Trial
Brief Title: Telemedicine for First Trimester Abortion in South Africa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Grand Challenges Canada (Other); University of California, San Francisco (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Deborah Constant, Dr, Director, Head of Women's Health Research Unit, Principal Investigator, Senior Researcher, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UCT HREC REF 671/2019
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Abortion in First Trimester
Keywords: Telemedicine screening; Eligibility for medical abortion; Improved access
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: inferiority randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Early medical abortion care (No Intervention): Counseling, history, instruction, family planning with clinic nurse. Ultrasound to assess gestational age.
- Telemedicine (Experimental): Online consultation questionnaire and counseling, family planning information. Instruction for the abortion received to the participants Facebook Messenger. Gestational age <9 weeks assessed by bimanual palpation, ultrasound only in case of uncertainty.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Telemedicine consultation online
  Arms: Telemedicine

SUMMARY:
The study aim to determine if medical abortion facilitated by a physician online (s.c. telemedicine), combined with a simplified physical exam, is equally effective, safe and acceptable to women in South Africa as standard medical abortion care.

DETAILED DESCRIPTION:
The proposed study is non-inferiority randomized controlled trial that will investigate the safety, effectiveness and acceptability for women of early medical abortion performed through telemedicine, compared to standard care in South Africa. Standard care, in the Western Cape, includes face to face eligibility screening, counselling and information with a nurse or physician, as well as an ultrasound to confirm the gestational age of the pelvic exam. The intervention will include a pelvic exam and gestatonal age based on LMP assessment and uterine size by bimanual palpation. Eligibility screening, counselling and information will occur through an existing online telemedicine application, content and language-adapted to suit women in South Africa, and managed by a HPCSA certified doctor. The study is a non-inferiority study. Our hypothesis is that the intervention is not inferior to standard care with respect to safety, effectiveness and acceptability. The study is performed to provide an alternate model of abortion care to be applied in settings where abortion is in any way restricted and increase access to safe abortion. Importantly the study is planned for a context where abortion services are legal but restricted by stigma. South Africa therefore provides a uniquely suited setting for this study.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write
* Able to speak English, IsiXhosa or Afrikaans
* Gestational age <9 wks 2 days
* In possession of a smartphone

Exclusion Criteria:

* Contraindication to medical abortion

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who took the abortion pills as instructed | 5 days after abortion consultation
  Proportion of women who successfully followed through with the abortion consultation and took the abortion pills as instructed
Rate of complete abortion. | 6 weeks after abortion consultation
  Effectiveness Rate of complete abortion. i.e. terminated pregnancy, without need of surgical or medical intervention or persistent bleeding within 6 weeks of the abortion initiation.

SECONDARY OUTCOMES:
Percentage of women visiting emergency hospital visit for abortion-related symptoms | 5 days after abortion consultation
  Emergency hospital visit for symptoms related to the abortion within two days of the intake of misoprostol
Percentage of women hospitalised for abortion complications | 5 days after abortion consultation
  Rate of hospitalization for complications to the abortion
Rate of blood transfusion for heavy bleeding | 5 days after abortion consultation
  Rate of blood transfusion for heavy bleeding during the abortion
Percentage of women preferring telemedicine to standard care | 6 weeks after abortion consultation
  Proportion of women selecting telemedicine vs standard care as a preferred option for a hypothetical future abortion
Proportion of women that were satisfied or very satisfied with their abortion consultation | 6 weeks after abortion consultation
  Proportion of women that were satisfied or very satisfied with their abortion consultation, telemedicine/standard care

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A CONSTANT, PhD, Principal Investigator — University of Cape Town
Locations (4):
- South Africa (4):
  - Karl Bremer Hospital, Bellville, Western Cape
  - Vanguard CHC, Cape Town, Western Cape
  - Michael Mapongwana CHC, Khayelitsha, Western Cape
  - Mitchells Plain CHC, Mitchells Plain, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Data base will be shared upon reasonable request accompanied by requester's protocol
Supporting Information: Study Protocol, ICF
Time Frame: After main findings have been published, for 3 years.
Access Criteria: Email request to Principal Investigators. Accompanied by requester's protocol and Ethics approval

REFERENCES:
- [Derived] Endler M, Petro G, Gemzell Danielsson K, Grossman D, Gomperts R, Weinryb M, Constant D. A telemedicine model for abortion in South Africa: a randomised, controlled, non-inferiority trial. Lancet. 2022 Aug 27;400(10353):670-679. doi: 10.1016/S0140-6736(22)01474-X. PMID 36030811